CLINICAL TRIAL: NCT06309940
Title: Prognostic Factors for Surgical Management of Large Hypertensive Basal Ganglionic Haemorrhage
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Sameeh, Resident doctor at neurosurgery Department, Assiut University
Other Study IDs: Basal ganglionic haemorrhage
Record Dates: First submitted 2024-03-07; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Basal Ganglionic Hemorrhage
MeSH Terms: conditions — Basal Ganglia Hemorrhage

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Prognostic factors of surgical evacuation of basal ganglionic haemorrhage — Surgical evacuation of basal ganglionic haemorrhage

SUMMARY:
The aim of this study is to present current and comprehensive recommendations for surgical treatment of this hematoma and to determine the factors that may improve the survival rate

DETAILED DESCRIPTION:
Spontaneous intracerebral hemorrhage is a common, mostly deadly stroke subtype and accounts for 10% to 15% of all strokes.

It's associated with a higher mortality rate (44% after 30 days) than either ischemic stroke or subarachnoid hemorrhage Up to 75% of the long term survivors are often suffering significant disability and only 12% to 39% of the survivors have favourable neurological functions recovered Rapid diagnosis and attentive management of patients is crucial because early deterioration is common Neurosurgical treatment for ICH has been discussed in recent multicentric studies, but no definitive answer of its utility has emerged.

Improved surgical techniques , neuroimaging, neuroanesthesia and perioperative monitoring and care have all led to improved outcomes from surgery

ELIGIBILITY:
Inclusion Criteria:

* 1) patients aged between 15 and 60 years old ( elderly people>60 years were excluded since their strokes weren't routinely examined by CT scan in the emergency ward, however, in children<15 years old was due mostly to vascular malformations 2) CT scan showed basal ganglionic haemorrhage, with or without intraventricular extension within 24 hr post ictus 3) hematoma volume was 30 ml or above 4) Glasgow Coma Scale scores more than or equal 5 and stable vital signs

Exclusion Criteria:

* 1) intracerebral hemorrhage was caused by secondary factors e.g ( vascular malformations or head trauma) 2) GCS less than 5 or multiple intracranial hemorrhage 3) associated visceral disease e.g hepatic or renal or clotting disorder 4) patients with preexisting neurological deficit e.g previous intracerebral hemorrhage or infarction

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Any adult patient of both sexes admitted to neurosurgery Department with non traumatic BG hemorrhage with total coverage of 1 year
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Prognostic factors of surgical evacuation of basal ganglionic haemorrhage | Baseline
  To investigate the effect of different factors on the outcome of the surgical evacuation of basal ganglionic haemorrhage

CONTACTS AND LOCATIONS:
Overall Officials: Farrag Mohamed, Doctor, Study Chair — Assiut University neurosurgery Department

REFERENCES:
- [Background] McCarron MO, Nicoll JA. Spontaneous intracerebral hemorrhage. N Engl J Med. 2001 Sep 6;345(10):769; author reply 770. doi: 10.1056/NEJM200109063451014. No abstract available. PMID 11547754
- [Background] Fernandes HM, Mendelow AD. Spontaneous intracerebral haemorrhage: a surgical dilemma. Br J Neurosurg. 1999 Aug;13(4):389-94. doi: 10.1080/02688699943501. PMID 10616566